CLINICAL TRIAL: NCT00287924
Title: Phase II Study of High-Dose Methotrexate in Children With Residual Ependymoma
Brief Title: High-Dose Methotrexate in Treating Young Patients With Residual Ependymoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454548; CCLG-CNS-2005-03; EU-20581; EUDRACT-2004-004405-14
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood infratentorial ependymoma; childhood supratentorial ependymoma; newly diagnosed childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Methotrexate; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: methotrexate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as methotrexate, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well high-dose methotrexate works in treating young patients with residual ependymoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the activity of high-dose methotrexate as upfront-window therapy in young patients with residual ependymoma.

Secondary

* Assess the reasons why primary surgery was complete/incomplete in these patients.
* Assess the feasibility and toxicity of second-look surgery after 3 courses of high-dose methotrexate in cases where initial surgery was incomplete.

OUTLINE: This is a multicenter, open-label study.

Patients receive high-dose methotrexate IV continuously over 24 hours on days 0, 14, and 28 in the absence of disease progression or unacceptable toxicity. Patients then proceed to further chemotherapy on protocol UKCCSG-CNS-9204.

After completion of study treatment, patients are followed periodically for 9 years.

PROJECTED ACCRUAL: A total of 29 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ependymoma, including the following histologic variants:

  * Cellular
  * Papillary
  * Clear-cell
  * Tanycytic
  * Anaplastic (malignant) ependymoma
* The following diagnoses are excluded:

  * Myxopapillary ependymoma
  * Subependymomas
  * Ependymoblastomas
  * Primitive neuroectodermal tumors (PNETs)
  * Other neuroepithelial tumors
  * Choroid plexus tumors
  * Germ cell tumors
* Residual measurable ependymoma after maximal surgical resection, including second-look surgery, if deemed necessary

  * Has undergone surgical resection within the past 3 weeks

PATIENT CHARACTERISTICS:

* At least 3 months to under 3 years of age
* Neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Able to tolerate chemotherapy
* No co-existent unrelated disease (i.e., renal or hematological) that would preclude chemotherapy treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior surgery
* No previous chemotherapy
* Previous steroids allowed
* No previous radiotherapy

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Estimated)
Dates: Start 2005-03; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Activity of high-dose methotrexate at 6 weeks

SECONDARY OUTCOMES:
Assess reasons why primary surgery is complete or incomplete at diagnosis
Feasibility and toxicity of second look surgery after course 3 at 2 months
Compare functional imaging studies of ependymomas with biological characteristics of the tumors at diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Martin W. English, MD, Study Chair — Birmingham Children's Hospital
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales